CLINICAL TRIAL: NCT01543763
Title: Phase I Study to Evaluate the Tolerability, Efficacy, and Safety of Pazopanib in Combination With PCI-24781 in Patients With Metastatic Solid Tumors
Brief Title: Pazopanib in Combination With PCI-24781 in Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pamela Munster (Other)
Collaborators: Pharmacyclics LLC. (Industry); Novartis (Industry); Xynomic Pharmaceuticals, Inc. (Industry); GlaxoSmithKline Research and Education Foundation for Cardiovascular Disease (Unknown)
Responsible Party: Sponsor-Investigator, Pamela Munster, Professor, Department of Medicine (Hematology/Oncology), UCSF, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11955; NCI-2012-01142 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-02-17; First posted 2012-03-05 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Solid Tumors
Keywords: metastatic; solid; sarcoma; progression
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Disease Progression | interventions — abexinostat; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Panobinostat with PC124871 (Experimental)
  Interventions: Drug: PZP115891, PCI-24781

INTERVENTIONS:
Drug: PZP115891, PCI-24781 — PCI-24781: oral, 30 to 75 mg/m2 b.i.d. Cycle 1, Days -7 to -4 and Cycle 1 and ongoing - Days 1-5, 8-12, 15-19
  PZP115891: oral, 400 - 800 mg qd 28 days per cycle
  Other Names: abexinostat; S 78454; GW786034; Votrient™; Pazopanib

SUMMARY:
This is a open-label non-randomized, dose escalation and expansion Phase Ia/Ib study to determine the safety, tolerability and maximum tolerated dose (MTD) of pazopanib in combination with PCI-24781 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Study rationale/purpose

Pazopanib is a potent, multi-targeted tyrosine kinase inhibitor44 of VEGFR-1, -2, -3, PDGFR-α and -β and c-kit approved for metastatic renal cell carcinoma based on phase III data showing a significant prolongation of progression-free survival (PFS) (5 mos in pretreated patients and 8.3 mos in treatment-naïve patients). In addition recent data was presented this year, but is not yet published, with treatment-refractory sarcoma patients that showed a PFS was significantly prolonged from a median of 20 vs. 7 weeks. As can occur with all antiangiogenic agents, resistance to pazopanib may develop. Epigenetic modification with HDAC inhibitors may overcome drug resistance by causing an increase in accessibility of DNA to chemotherapeutic agents and may therefore significantly potentiate their cytotoxicity. Combination trials with chemotherapy agents are ongoing (ClinicalTrials.gov) To our knowledge, a combination trial of HDACi with anti-angiogenesis agents has not yet been performed and represents an unmet medical need.

PCI-24781 is a pan HDAC inhibitor. In cell lines tested, up-regulation and down-regulation of genes known to result in changes with signal transduction, oxidation, metabolic changes, apoptosis, proliferation, differentiation and angiogenesis were seen. In addition, ongoing single agent and combination trials have shown the drug to be effective and well-tolerated.

Hypothesis: Combining an antiangiogenic agent, such as pazopanib, with an epigenetic modifier, such as histone deacetylase inhibitor (HDACi) PCI-24781, can increase the efficacy of pazopanib as well as overcome development of resistance to pazopanib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to adhere with treatment and followup.
2. Age ≥ 18 years
3. Phase Ia: Patients must have histologically or cytologically documented metastatic solid tumor malignancies. Phase Ib: Patients must have histologically or cytologically confirmed locally advanced, solid tumor malignancies of one of the following tumor types:

   1. Renal cell carcinoma (N = 20 patients) (Cohort A)
   2. Non-anaplastic thyroid carcinoma (N = 20 patients) (Cohort B) Documentation of histology from a primary or metastatic site is allowed.
   3. Soft tissue sarcoma (N = 20 patients) (Cohort C). Patients must have progressed in a prior line of therapy.
   4. Ovarian carcinoma (N = 20 patients) (Cohort D)
4. Measurable disease by RECIST 1.1
5. Phase Ia: Patients may have de novo metastatic disease, or documented progression despite any number of prior therapies. Patients must have no curative or other effective therapeutic options available. Phase Ib: Patients may have had any number of prior treatments, or prior pazopanib.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
7. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower except for alopecia
8. Patient must be at least 4 weeks or five half-lives (whichever is shorter) from last standard or experimental therapy, except Patients who have received prior pazopanib are eligible but must not have received it in the last two weeks.
9. Patients must be at least 28 days from last radiation therapy dose, Peptide Receptor Radionuclide Therapy (PRRT), surgery, or tumor embolization prior to the first dose of pazopanib/PCI-24781
10. A female is eligible to enter and participate in this study if she is of:

    1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

       * A hysterectomy
       * A bilateral oophorectomy (ovariectomy)
       * A bilateral tubal ligation
       * Is post-menopausal Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, or, in questionable cases, have a follicle stimulating hormone (FSH) value >40 milli-international units per millilitre (mIU/mL) and an estradiol value < 40pg/mL (<140 pmol/L). Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
    2. Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Novartis Pharmaceuticals acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

       * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
       * Oral contraceptive, either combined or progestogen alone
       * Injectable progestogen
       * Estrogenic vaginal ring
       * Percutaneous contraceptive patches
       * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
       * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
       * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
       * Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
11. Adequate organ system function as defined below

    * Absolute neutrophil count (ANC) 1.5 X 109/L
    * Hemoglobin 9 g/dL (5.6 mmol/L)
    * Platelets 100 X 109/L
    * Prothrombin time (PT) or international normalized ratio (INR) 1.2 X upper limit of normal (ULN)
    * Activated partial thromboplastin time (aPTT) 1.2 X ULN
    * Total bilirubin 1.5 X ULN
    * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) 2.5 X ULN
    * Serum creatinine <1.5 x ULN Or, if >1.5 mg/dL: Calculated creatinine clearance 50 mL/min Urine Protein to Creatinine Ratio (UPC) e <1
12. Subjects may not have had a transfusion within 7 days of screening assessment.
13. Subjects receiving anticoagulant therapy are eligible if their INR is within the recommended range for the desired level of anticoagulation.
14. Patients with increased bilirubin due to Gilberts disease will not be excluded, if increased bilirubin is the only protocol exclusion criteria met.
15. Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.
16. If UPC ≥1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 g to be eligible.

5.1.2 Exclusion Criteria

1. Patients with other primary malignancies receiving active treatment at the time of study entry, other than carcinoma in situ of the cervix, non-melanoma skin cancer, nonmuscle invasive bladder cancer.
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
4. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   * Malabsorption syndrome
   * Major resection of the stomach or small bowel.
5. Presence of known active hepatitis C viral (HCV) or active hepatitis B viral (HBV) infection, history of human immunodeficiency virus (HIV), or other uncontrolled systemic infection
6. Corrected QT interval (QTc) > 480 msecs using Bazett's formula
7. Concurrent use of medications that are known to prolong or cause QT prolongation
8. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
9. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA), see Appendix A
10. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥160 mmHg or diastolic blood pressure (DBP) of ≥ 100 (mmHg].

    Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) Systolic Blood Pressure/Diastolic Blood Pressure values from each blood pressure assessment must be <160/100 mmHg in order for a subject to be eligible for the study.
11. History of cerebrovascular accident, including transient ischemic attack (TIA)
12. History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months Note: Patients with recent DVT who have been treated with therapeutic anticoagulation including Coumadin or any low molecular weight heparin for at least 6 weeks are eligible
13. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
14. Evidence of active bleeding or bleeding diathesis
15. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedures
16. Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is shorter) prior to the first dose of study drug and for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 4 weeks
  A dose limiting toxicity (DLT) will be defined as any predetermined adverse events occurring during Cycle 1 when association to therapy that is part of this study is related or possibly related
Maximum Tolerated Dose (MTD) | up to 4 weeks
  The maximum tolerated dose (MTD) will be defined as the highest tested dose level at which less than 33% of patients experience DLT in Cycle 1

SECONDARY OUTCOMES:
Establish the volume of distribution of PCI-24781, pazopanib and the combination of the two drugs. | up to 2 months
  Noncompartmental pharmacokinetic profile of PCI-24781, pazopanib and the combination will be assessed by measuring and calculating the volume of distribution (Vd)
Establish the bioavailability of PCI-24781, pazopanib and the combination of the two drugs. | up to 2 months
  Noncompartmental pharmacokinetic profile of PCI-24781, pazopanib and the combination will be assessed by measuring and calculating the bioavailability (F).
Establish the clearance of PCI-24781, pazopanib and the combination of the two drugs. | up to 2 months
  Noncompartmental pharmacokinetic profile of PCI-24781, pazopanib and the combination will be assessed by measuring and calculating clearance (CL)
Establish the half-life of PCI-24781, pazopanib and the combination of the two drugs. | up to 2 months
  Noncompartmental pharmacokinetic profile of PCI-24781, pazopanib and the combination will be assessed by measuring and calculating the half-life (t1/2)
Establish the area under the curve (AUC) of PCI-24781, pazopanib and the combination of the two drugs. | up to 2 months
  Noncompartmental pharmacokinetic profile of PCI-24781, pazopanib and the combination will be assessed by measuring and calculating the AUC
Clinical Benefit Rate (CBR) | approximately 4 months
  Clinical Benefit Rate=Complete Response (CR)+Partial Response (PR)+Stable Disease (SD) is defined as the best response at any time or maintaining stable disease for at least 12 weeks and will be evaluated by imaging criteria RECIST 1.1. A patient with unknown or missing response will be treated as a non-responder. Patients are expected to receive treatment for at least 2 Cycles, at which time the first evaluation for efficacy will occur. Exact methods for calculated confidence intervals will be utilized.
Objective response rate (ORR) | approximately 4 months
  Objective response rate is defined as the percentage or proportion of patients with a confirmed complete or partial response (CR+PR) as defined by RECIST 1.1 divided by the total number of patients on study. Patients are expected to receive treatment for at least 2 Cycles, at which time the first evaluation for efficacy will occur. A patient with unknown or missing response will be treated as a non-responder. Exact methods for calculated confidence intervals will be utilized.
Progression-free Survival (PFS) | Up to 1 year
  Time to progression will be calculated as the time from first dose of the combination until the earliest date of documented disease relapse, progression, or death from any cause. If the patient does not have a documented date of progression or death, then PFS will be censored at the date of last adequate assessment. PFS will be summarized using Kaplan-Meier method and lifetables, including the 1-year point estimates with standard errors.
Overall survival (OS) | Up to 1 year
  Overall survival will be calculated as the time from first dose of the combination until the earliest date of documented study discontinuation or death from any cause. If the patient does not have a documented date of death, then OS will be censored at the date of last adequate assessment. OS will be summarized using Kaplan-Meier method and lifetables, including the 1-year point estimates with standard errors.
Duration of Response (DoR) | Up to 1 year
  Duration of Response is defined, for the subset of patients with a confirmed complete or partial response, as the time from first documented evidence of CR or PR until first documented disease progression or death due to any cause. Only the subset of patients who show a confirmed complete or partial tumor response will be included. Censoring rules for duration of response will follow the rules for PFS

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No